CLINICAL TRIAL: NCT00763503
Title: Pharmacokinetic and Pharmacodynamic Study of CD 2027 3µg/g Oily Spray Applied Twice Daily for 3 Weeks Under Conditions of Maximized Use in Adults With Plaque-type Psoriasis
Brief Title: Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of CD 2027 Spray in Adults With Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18118
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2012-01

CONDITIONS: Plaque-type Psoriasis
Keywords: psoriasis; PK; calcitriol
MeSH Terms: conditions — Psoriasis | interventions — Calcitriol

ARMS (1):
- CD 2027 (Experimental)
  Interventions: Drug: CD 2027

INTERVENTIONS:
Drug: CD 2027 — 3µg/g Oily Spray
  Other Names: Calcitriol

SUMMARY:
This is a multicenter, open-label study to assess systemic plasma levels of calcitriol, calcium homeostasis and safety in adults with plaque-type psoriasis under conditions of maximized use of CD 2027 3µg/g oily spray twice daily (6 g daily), applied to 20% of BSA for 3 weeks.

There are a total of six visits: Pre-treatment period (Day -15, Day -8 and Day -1) and Treatment period (Day 1/ Baseline, Day 15 and Day 22).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque-type psoriasis involving 10% - 20% of body surface area (BSA), with a Global Severity Score of at least 3 (moderate)

Exclusion Criteria:

* Other type of psoriasis (other than plaque)
* Significant abnormal lab findings
* Secondary hyperparathyroidism
* Vit D deficiency
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
CD 2027 plasma concentrations | 0, 1, 2, 3, 4, 6, 9, 12 hour time points

SECONDARY OUTCOMES:
Calcium homeostasis | Screening, Day -8, -1 and prior to the morning application on Day 1, 15 and 22

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - DermResearch, Austin, Texas
  - J & S Studies, Bryan, Texas